CLINICAL TRIAL: NCT03620006
Title: Endovascular Occlusion by Plug of the Prevertebral Subclavian Artery Preparatory to the Surgical or Endovascular Aortic Procedures (SAPE)
Brief Title: Subclavian Artery Plug Embolization (SAPE)
Acronym: SAPE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: SAPE
Record Dates: First submitted 2018-05-21; First posted 2018-08-08 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Subclavian Artery Plug Embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, no-profit, ambispective study: a retrospective arm will include the cases treated between August 2009 and March 2018, and a prospective arm, investigating patients treated from March 2018 until December 2018. Target study population size is 150 patients between two groups analyzed.

Endovascular occlusion of the prevertebral subclavian artery was first used in the Vascular Surgery Department at San Raffaele Hospital in August 2009. During the initial experience (2009-2014) this technique was used with low frequency. Since 2015, the volume of cases receiving this treatment, has increased and the investigators expect to reach the study population target, by the end of 2018.

The objective of this study is describe the casuistry of endovascular occlusion of the subclavian artery by means of the Amplatzer Vascular plug in the Vascular Surgery Department at San Raffaele Hospital, and to evaluate the efficacy of such procedure.

Moreover, the investigators will evaluate the patency and success rate of the carotid-subclavian bypasses performed at the same time of the analyzed procedure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged ≥ 18 years,
* patients candidates for endovascular treatment of subclavian artery occlusion with Amplatzer Vascular Plug

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients aged ≥ 18 years, candidates for endovascular treatment of subclavian artery occlusion with Amplatzer Vascular Plug
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Technical success rate | within 30-day
  Technical success rate defined as complete occlusion of the left subclavian artery at postoperative CT scan
Major adverse event rate | within 30-day
  Any stroke or mortality related to the surgical procedure

SECONDARY OUTCOMES:
Access site complications requiring secondary adjunctive procedures | within 30-day
  Any access site complication requiring open or endovascular adjuctive procedures (ie: surgical embolectomy, echo-guided pseudoaneurysm manual compression)
Supra-aortic vessels patency rate | within 5-years
  Patency of the carotid and subaclavian artery at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertoglio L, Salvati S, Fittipaldi A, Melloni A, Kahlberg A, Cambiaghi T, Melissano G, Chiesa R. Carotid to subclavian bypass and Amplatzer vascular plug subclavian endovascular occlusion before thoracic open or endovascular repair. J Vasc Surg. 2020 May;71(5):1480-1488.e1. doi: 10.1016/j.jvs.2019.08.237. Epub 2019 Oct 17. PMID 31630886